CLINICAL TRIAL: NCT03630224
Title: Renal Effects of Fluid Resuscitation With Plasmalyte Viaflo Versus Saline in Trauma Patients (the ASTRAU Study)
Brief Title: Plasmalyte Versus Saline in Trauma Patients
Acronym: ASTRAU
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Premature termination due to futility following interim analysis
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P160919J; 2017-004206-17 (Other: IDRCB)
Record Dates: First submitted 2018-08-10; First posted 2018-08-14 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Severe Trauma Patients; Acute Kidney Injury
Keywords: Severe trauma; Acute kidney injury; Fluid resuscitation; Sodium chloride; Plasmalyte
MeSH Terms: conditions — Acute Kidney Injury; Wounds and Injuries | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plasmalyte Viaflo (Experimental): Intervention type: drug (Plasmalyte Viaflo) Intervention name: plasmalyte Intervention description: fluid resuscitation using exclusively Plasmalyte up to 20L during the first 5 days
  Interventions: Drug: Plasmalyte Viaflo
- NaCl 0.9% (Active Comparator): Intervention type: drug (NaCl 0.9%) Intervention name: NaCl 0.9% Intervention description: fluid resuscitation using exclusively NaCl 0.9% up to 20L during the first 5 days
  Interventions: Drug: NaCl 0.9%

INTERVENTIONS:
Drug: Plasmalyte Viaflo — Intervention description: fluid resuscitation using exclusively Plasmalyte up to 20L during the first 5 days
  Arms: Plasmalyte Viaflo
Drug: NaCl 0.9% — Intervention name: NaCl 0.9% Intervention description: fluid resuscitation using exclusively NaCl 0.9% up to 20L during the first 5 days
  Arms: NaCl 0.9%

SUMMARY:
Fluid resuscitation remains the cornerstone for the care of severe trauma patients to compensate for blood loss, to compensate for capillary leak induced by systemic inflammation but also to prevent the detrimental consequences of traumatic rhabdomyolysis. Isotonic saline (NaCl 0.9%), called "physiological serum" is the standard fluid for the resuscitation of severely injured patients. However, the formulation of NaCl 0.9% is not really physiological since its chloride concentration is 1.5 higher than the one of human plasma. This excessive chloride concentration leads to hyperchloremic acidosis and to a drop in renal perfusion after isotonic saline infusion. For this reason, we wonder whether fluid resuscitation with Plasmalyte would be beneficial for renal function of trauma patients in comparison with NaCl 0.9%. Our research question is:

In a population of trauma patients at high risk of acute kidney injury, does a fluid resuscitation with Plasmalyte Viaflo lower the incidence of severe acute kidney injury (stage 2 or 3 according to the KDIGO classification) compared with a resuscitation with isotonic saline (NaCl 0.9%)?

DETAILED DESCRIPTION:
Fluid resuscitation remains the cornerstone for the care of severe trauma patients to compensate for blood loss, to compensate for capillary leak induced by systemic inflammation but also to prevent the detrimental consequences of traumatic rhabdomyolysis. Isotonic saline (NaCl 0.9%), called "physiological serum" is the standard fluid for the resuscitation of severely injured patients. However, the formulation of NaCl 0.9% is not really physiological since its chloride concentration is 1.5 higher than plasma. This excessive chloride concentration leads to hyperchloremic acidosis and to a drop in renal perfusion after isotonic saline infusion. A retrospective study conducted in the perioperative setting (abdominal surgery) reported a significant decrease in mortality and acute kidney injury in 926 patients receiving balanced crystalloid solution compared to a propensity-matched population of 2778 patients receiving isotonic saline. Yunos et al. conducted a prospective sequential period study including 760 patients receiving chloride-rich solution during the first 6-month period and 773 patients receiving chloride-poor solution during the next 6-month period. They reported a decrease in severe acute kidney injury (I or F in the RIFLE classification) in the group receiving chloride-poor solution. Large retrospective studies in intensive care confirmed a beneficial effect of the use of chloride-poor solutions on survival compared to chloride-rich solutions. A recent meta-analysis including 5 small size randomized controlled trials, 1 controlled trial and two retrospective studies, reported also a decrease in acute kidney injury. A recent multicenter study randomized 2778 patients to receive either Plasmalyte 148 or NaCl 0.9% during their ICU stay. No AKI or mortality differences were reported. However, this study included patients with low ICU severity score (mean APACHE II = 14) and at low risk of severe AKI (severe AKI incidence = 9%). Moreover, they received a median amount of fluid of 2000 mL during their ICU stay. This small fluid volume may not be enough to show any difference between rich-chloride and poor-chloride solutions on AKI in this population with low ICU severity scores.

Trauma patients are particularly at risk of AKI during the acute phase of trauma because of hypovolemia (bleeding), rhabdomyolysis and systemic inflammation (traumatic tissue injuries and emergency surgeries). AKI is reported in 18 to 26 % of trauma patients. In our database (TraumaBase®, traumabase.eu) that included at the time of the study the 6 trauma centers of the Paris area (France), we reported a 24% incidence of severe AKI (stage I or F of the RIFLE classification) in the subpopulation of patients needing at least one red blood cell unit transfusion in the 6 first hours of care. Moreover, this subpopulation receives an average amount of 6000 mL of fluid during the first 24 hours of care. We postulate that trauma patients at high risk of AKI receiving high volume of fluid can be the best population target to demonstrate a beneficial effect of Plasmalyte vs isotonic saline on severe AKI occurrence in a prospective, blinded, randomized manner.

Thus, we formulate the following hypothesis:

In a population of trauma patients, at high risk of AKI, a fluid resuscitation with Plasmalyte Viaflo during the 5 first days of care will lower decrease the incidence of severe acute kidney injury (stage 2 or 3 according to the KDIGO classification) compared with a resuscitation with isotonic saline (NaCl 0.9%)

ELIGIBILITY:
Inclusion Criteria:

* Severe trauma defined by at least one Vittel criteria
* Prescription for at least one red blood cell unit transfusion within 6 hours after trauma
* Delay between trauma and study randomization ≤ 6 hours
* Patient able to give consent or included in emergency situation
* Patient affiliated to Health security system

Exclusion Criteria:

* Age < 18 years
* Chronic kidney disease needing requiring renal replacement therapy
* Participation to another interventional trial interacting with renal function or which requires the use of a fluid resuscitation
* Fluid resuscitation > 4000 mL before inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-08-18 (Actual)

PRIMARY OUTCOMES:
Proportion of Acute Kidney Injury (stage 2 or 3 according to KDIGO classification) over the 5 first days after trauma | over the 5 first days after trauma

SECONDARY OUTCOMES:
Proportion of patients requiring renal replacement therapy (during 28 days) | during 28 days
Amount of transfused blood product units (during the first 5 days) | during the first 5 days
Number of days alive without free of mechanical ventilation (during 28 days) | during 28 days
Days spent alive outside the ICU (during 28 days) | during 28 days
Mortality | at 28 days
Difference between the serum creatinine peak in the 5 first days of ICU stay and the baseline creatinine | during the 5 first days

CONTACTS AND LOCATIONS:
Overall Officials: Anatole HARROIS, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Département d'Anesthésie Réanimation - Kremlin Bicêtre, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chowdhury AH, Cox EF, Francis ST, Lobo DN. A randomized, controlled, double-blind crossover study on the effects of 2-L infusions of 0.9% saline and plasma-lyte(R) 148 on renal blood flow velocity and renal cortical tissue perfusion in healthy volunteers. Ann Surg. 2012 Jul;256(1):18-24. doi: 10.1097/SLA.0b013e318256be72. PMID 22580944
- [Background] Shaw AD, Bagshaw SM, Goldstein SL, Scherer LA, Duan M, Schermer CR, Kellum JA. Major complications, mortality, and resource utilization after open abdominal surgery: 0.9% saline compared to Plasma-Lyte. Ann Surg. 2012 May;255(5):821-9. doi: 10.1097/SLA.0b013e31825074f5. PMID 22470070
- [Background] Yunos NM, Bellomo R, Hegarty C, Story D, Ho L, Bailey M. Association between a chloride-liberal vs chloride-restrictive intravenous fluid administration strategy and kidney injury in critically ill adults. JAMA. 2012 Oct 17;308(15):1566-72. doi: 10.1001/jama.2012.13356. PMID 23073953
- [Background] Shaw AD, Raghunathan K, Peyerl FW, Munson SH, Paluszkiewicz SM, Schermer CR. Association between intravenous chloride load during resuscitation and in-hospital mortality among patients with SIRS. Intensive Care Med. 2014 Dec;40(12):1897-905. doi: 10.1007/s00134-014-3505-3. Epub 2014 Oct 8. PMID 25293535
- [Background] Raghunathan K, Shaw A, Nathanson B, Sturmer T, Brookhart A, Stefan MS, Setoguchi S, Beadles C, Lindenauer PK. Association between the choice of IV crystalloid and in-hospital mortality among critically ill adults with sepsis*. Crit Care Med. 2014 Jul;42(7):1585-91. doi: 10.1097/CCM.0000000000000305. PMID 24674927
- [Background] Shaw AD, Schermer CR, Lobo DN, Munson SH, Khangulov V, Hayashida DK, Kellum JA. Impact of intravenous fluid composition on outcomes in patients with systemic inflammatory response syndrome. Crit Care. 2015 Sep 12;19(1):334. doi: 10.1186/s13054-015-1045-z. PMID 26370823
- [Background] Krajewski ML, Raghunathan K, Paluszkiewicz SM, Schermer CR, Shaw AD. Meta-analysis of high- versus low-chloride content in perioperative and critical care fluid resuscitation. Br J Surg. 2015 Jan;102(1):24-36. doi: 10.1002/bjs.9651. Epub 2014 Oct 30. PMID 25357011
- [Background] Young P, Bailey M, Beasley R, Henderson S, Mackle D, McArthur C, McGuinness S, Mehrtens J, Myburgh J, Psirides A, Reddy S, Bellomo R; SPLIT Investigators; ANZICS CTG. Effect of a Buffered Crystalloid Solution vs Saline on Acute Kidney Injury Among Patients in the Intensive Care Unit: The SPLIT Randomized Clinical Trial. JAMA. 2015 Oct 27;314(16):1701-10. doi: 10.1001/jama.2015.12334. PMID 26444692
- [Background] Bagshaw SM, George C, Gibney RT, Bellomo R. A multi-center evaluation of early acute kidney injury in critically ill trauma patients. Ren Fail. 2008;30(6):581-9. doi: 10.1080/08860220802134649. PMID 18661407
- [Background] Bihorac A, Delano MJ, Schold JD, Lopez MC, Nathens AB, Maier RV, Layon AJ, Baker HV, Moldawer LL. Incidence, clinical predictors, genomics, and outcome of acute kidney injury among trauma patients. Ann Surg. 2010 Jul;252(1):158-65. doi: 10.1097/SLA.0b013e3181deb6bc. PMID 20562612